CLINICAL TRIAL: NCT00000442
Title: Etiology and Treatment of Alcohol Dependence
Brief Title: Naltrexone for Relapse Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Henry Kranzler, University of Pennsylvania
Model: Parallel | Purpose: Treatment
Other Study IDs: NIAAAKRA3510; P50AA003510 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

INTERVENTIONS:
Drug: naltrexone (Revia)

SUMMARY:
This study is to evaluate the safety and effectiveness of an injectable slow releasing preparation of naltrexone to reduce alcohol consumption and risk of relapse in alcohol-dependent subjects. Individuals will receive either naltrexone or a placebo injection for a total of three months, with two subsequent followup visits spanning a 6- month period.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence.
* Abstinent from alcohol for a period of at least 3 days prior to beginning of study.
* Able to read English and complete study evaluations.
* Females who are postmenopausal, have had surgical sterilization, or use reliable means of birth control.

Exclusion Criteria:

* Meets criteria for dependence on a psychoactive substance other than alcohol and nicotine and/or cannabis.
* Prior history of opioid dependence.
* Regular use of psychoactive drugs including anxiolytics and antidepressants.
* Prior treatment with naltrexone.
* Current use of disulfiram.
* Psychotic or otherwise severely psychiatrically disabled (e.g., suicidal, current mania).
* Significant underlying medical conditions such as hepatic, cerebral, renal, thyroid, or cardiac disease.
* Abstinent longer than 28 days prior to randomization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57
Dates: Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania, United States